CLINICAL TRIAL: NCT02569320
Title: A Phase 1b Trial of AR-42 With Pomalidomide in Relapsed Multiple Myeloma
Brief Title: HDAC Inhibitor AR-42 and Pomalidomide in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-15004; NCI-2015-01557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PO-CL-MM-PI-003687
Record Dates: First submitted 2015-10-03; First posted 2015-10-06 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; HDAC-42; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pomalidomide, dexamethasone, HDAC inhibitor AR-42) (Experimental): Patients receive pomalidomide PO daily on days 1-21, dexamethasone PO BIW or TIW weeks 1-3, and HDAC inhibitor AR-42 PO BIW or TIW for weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: HDAC Inhibitor AR-42; Other: Laboratory Biomarker Analysis; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: HDAC Inhibitor AR-42 — Given PO
  Other Names: AR-42; HDAC-42; OSU-HDAC42
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Pomalyst

SUMMARY:
This pilot phase I trial studies the side effects and best dose of histone deacetylase (HDAC) inhibitor AR-42 (AR-42) when given together with pomalidomide in treating patients with multiple myeloma that has returned after a period of improvement. HDAC inhibitor AR-42 may work to stop cancer growth by blocking an enzyme needed for cell growth. Pomalidomide is a drug used in chemotherapy that works to stop the growth of cancer cells by causing them to die. Giving HDAC inhibitor AR-42 together with pomalidomide may cause patients to respond better to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose, safety and efficacy of AR-42 in combination with pomalidomide in relapsed multiple myeloma (MM) patients.

SECONDARY OBJECTIVES:

I. To determine time to progression (TTP). II. To determine overall survival (OS).

OUTLINE: This is a dose-escalation study of HDAC inhibitor AR-42 and pomalidomide.

Patients receive pomalidomide orally (PO) daily on days 1-21, dexamethasone PO twice weekly (BIW) or thrice weekly (TIW) weeks 1-3, and HDAC inhibitor AR-42 PO BIW or TIW on weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable disease as defined by any of the following:

  * Serum M-protein >= 0.5 g/dl (>= 500 mg/dL)
  * Urine monoclonal protein >= 200 mg/24h
  * Involved free light chain (FLC) level >= 10 mg/dl (>= 100 mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
* Patients must have previously received Lenalidomide and proteasome inhibitor.
* Patients must be lenalidomide failures: disease progression on a prior lenalidomide-based therapy or progression within 60 days of the last dose of a lenalidomide; patients should have received at least 2 cycles of a lenalidomide-based regimen at standard doses to be evaluable for refractoriness; prior intolerance to lenalidomide does not exclude participation in the study except in cases of severe allergic reaction
* Prior radiation is permitted; however, at least 2 weeks must have elapsed since the completion of therapy and patients must have recovered from all therapy-associated toxicities to no greater than grade 1 at the time of registration; patients with symptomatic disease may receive palliative corticosteroids up to 1 week before initiating therapy
* Patient must have received 2 or more prior lines of systemic therapy for myeloma; patients must be off last treatment for at least 2 weeks (wks) by the beginning of treatment on this protocol
* Patients must have a Karnofsky performance score of 50% or greater
* Patients must have absolute neutrophil count (ANC) > 1000/uL
* Platelets >= 75,000/uL
* Total bilirubin =< 1.5 mg/dL
* Alkaline phosphatase =< 4 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x IULN
* Patients must have a serum creatinine limit of ≤1.5 ULN or creatinine clearance of ≥60 ml/min measured within 14 days of registration.
* All study participants must be registered into the mandatory POMALYST (pomalidomide) Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the POMALYST REMS program
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL prior to starting therapy and prior to beginning another cycle (if applicable); women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* The patient must be willing to comply with fertility requirements as below:

  * Male patients must agree to use an adequate method of contraception for the duration of the study and for 28 days afterwards
  * Female patients must be either postmenopausal, free from menses >= 2 yrs, surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from heterosexual activity starting with screening (4 weeks prior to initiating treatment) and 28 days after treatment, per POMALYST REMS™ program
  * Patients must agree not to donate blood, sperm/ova during the course of taking protocol therapy and for at least 4 weeks after stopping treatment

Exclusion Criteria:

* History of severe allergic reaction, including erythema nodosum, to lenalidomide
* Patients unable to receive adequate thromboprophylaxis in combination with pomalidomide
* Patients who have received investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Patients with a mean QT interval corrected by Bazett's formula (QTcB) > 450 msec in males and > 470 msec in females
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C
* Patients with active (untreated or relapsed) central nervous system (CNS) metastasis of the patient's myeloma
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* Patients with a prior history of malignancies, other than multiple myeloma, are excluded unless the subject has been free of the disease for ≥ 5 years with the exception of the following non-invasive malignancies:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histological finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative.
* Patients with malabsorption or any other condition that in the opinion of the principal investigator could cause difficulty in absorption of drug
* Patients that have previously progressed on pomalidomide treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HDAC inhibitor AR-42 in combination with pomalidomide, defined as the highest dose level at which less than 20% of patients experience a dose-limiting toxicity | 21 days
  In the scenario where the MTD does not follow the assumption of non-decreasing toxicity of dose in both directions of the agent dose combinations, the MTD will be estimated by a bivariate isotonic estimator.

SECONDARY OUTCOMES:
Change in biomarker levels | Baseline to up to 30 days after completion of study treatment
  Summary statistics will be computed for baseline biomarkers. The absolute and percent change from baseline will be calculated for each subsequent measurement. Summary statistics will be computed for each collection time point.
Clinical benefit, defined as the proportion of patients experiencing complete response, very good partial response, or partial response | Up to 30 days after completion of study treatment
Duration of response | From first observation of partial response to the time of disease progression (taking as a reference for progressive disease the smallest measurements recorded since treatment started), assessed up to 30 days after completion of study treatment
  Evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.
Incidence of toxicity, evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4 standard toxicity grading | Up to 30 days after completion of study treatment
  Frequency distributions and other descriptive measures will form the basis of analysis of toxicity number and severity. Adverse events will be summarized by CTCAE v.4 category and perceived causal relationship to the study therapy. Tolerability will also be determined through assessing the number of patients who required dose modifications and/or dose delays in subsequent cycles. In addition, the proportion of patients who go off treatment due to adverse reactions or those who refuse further treatment for lesser toxicities that inhibit their willingness to continue on trial will be captured.
Number of patients experiencing objective response, based on criteria adapted from the International Myeloma working Group Uniform Response Criteria | Up to 30 days after completion of study treatment
  The number and percentage of patients experiencing objective response will be descriptively summarized overall and by dose level. The objective response rate will be analyzed by using a 95% confidence interval for the proportion responding at trial closure in the treated population.
Progression-free survival | From start of treatment to disease progression or death, regardless of cause of death, whichever comes first, assessed up to 30 days after completion of study treatment
  Evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.
Time to progression | From the start of the treatment until the criteria for disease progression are met, assessed up to 30 days after completion of study treatment
  Evaluated using the methods of Kaplan and Meier, with a focus on graphical evaluation as well as early timepoint and median estimates of survival distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Efebera, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng H, Xie Z, Jones WP, Wei XT, Liu Z, Wang D, Kulp SK, Wang J, Coss CC, Chen CS, Marcucci G, Garzon R, Covey JM, Phelps MA, Chan KK. Preclinical Pharmacokinetics Study of R- and S-Enantiomers of the Histone Deacetylase Inhibitor, AR-42 (NSC 731438), in Rodents. AAPS J. 2016 May;18(3):737-45. doi: 10.1208/s12248-016-9876-3. Epub 2016 Mar 4. PMID 26943915
- See also: The Jamesline — http://cancer.osu.edu